CLINICAL TRIAL: NCT05563909
Title: Investigation of the Efficacy of Virtual Reality Mediated Neurodynamic Exercises in Carpal Tunnel Syndrome: A Prospective Randomized Controlled Clinical Study
Brief Title: Investigation of the Efficacy of Virtual Reality Mediated Neurodynamic Exercises in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ahmet Kivanc Menekseoglu, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 07/09/2020-142688
Record Dates: First submitted 2022-09-24; First posted 2022-10-03 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 54 patients with CTS who met the inclusion criteria will be included in this prospectively planned study. At the beginning of the study, 54 patients with a diagnosis of CTS who met the inclusion criteria will be randomized into three groups according to the random order created by a computer program after being numbered according to the general polyclinic application order of Istanbul University, Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation.
Who Masked: Outcomes Assessor
Masking Description: The researcher evaluating the participants will be blind to the group distributions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Group (Experimental): Tendon and nerve gliding exercises will be applied to the patients in the virtual reality group for 2 weeks, for a total of 10 sessions, through the developed software. Patients will be asked to come for 2 weeks for the virtual reality mediated exercise program. Patients will be asked to do their exercises in a virtual reality-mediated exercise protocol, with 1 session of approximately 30 minutes. Apart from the exercise program, patients will be asked to use wrist splints.
  Interventions: Other: Wrist Splint; Other: Virtual Reality Mediated Exercise
- Conventional Exercise Group (Active Comparator): For the patients in the classical exercise group; The classical exercise program will be taught in the company of a physiotherapist and they will be asked to do these exercises for a total of 10 sessions for 2 weeks. The patients' home exercise programs will be controlled by weekly phone calls. Apart from the exercise program, patients will be asked to use wrist splints.
  Interventions: Other: Exercise; Other: Wrist Splint
- Control Group (Active Comparator): Patients in the control group will be advised to continue using splints. It will be evaluated by repeated examinations.
  Interventions: Other: Wrist Splint

INTERVENTIONS:
Other: Exercise — Patients participating in the study will not receive any intervention other than exercise and splint.
  Arms: Conventional Exercise Group
Other: Wrist Splint — Patients participating in the study will not receive any intervention other than exercise and splint.
Other: Virtual Reality Mediated Exercise — Patients participating in the study will not receive any intervention other than exercise and splint.
  Arms: Virtual Reality Group

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common nerve entrapment syndrome. It occurs as a result of compression of the median nerve as it passes through a restricted osteofibrous canal in the wrist. Known as the carpal tunnel, this canal contains the wrist bones, transverse carpal ligament, median nerve, and digital flexor tendons. Edema, tendon inflammation, hormonal changes, and manual activity can contribute to increased nerve compression and sometimes cause pain.

In this research, the investigators aim to present the virtual reality-mediated exercise program to patients non-immersive. It is planned to use the Leap Motion motion sensor to detect hand and wrist movements and to monitor the gamified setup on the computer screen.

In the system that will be presented via computer and hand motion sensor, the patient will be asked to perform therapeutic exercises for the diagnosis of CTS in a scenario developed through virtual reality. The investigators predict that patients will actively participate in virtual reality-mediated therapeutic exercise program with high motivation and their functional results will be better than classical exercise programs.

In our research, the investigators aim to present the tendon and nerve gliding exercises with proven effectiveness in patients with CTS, with non-immersive virtual reality systems, and to compare their effectiveness with the classical exercise program.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common nerve entrapment syndrome. It occurs as a result of compression of the median nerve as it passes through a restricted osteofibrous canal in the wrist. Known as the carpal tunnel, this canal contains the wrist bones, transverse carpal ligament, median nerve, and digital flexor tendons. Edema, tendon inflammation, hormonal changes, and manual activity can contribute to increased nerve compression and sometimes cause pain. In more severe cases, weakness may occur in the muscles innervated by the median nerve, resulting in weakness in hand muscle strength(1). In a comprehensive study, the mean age for the diagnosis of CTS was found to be 50 years, and its prevalence was found to be similar in men and women. However, the prevalence was higher in women; The incidence in women aged 65-74 was found to be four times higher than in men(2).

Many different treatment methods are used in the treatment of CTS, and these treatments include regulation of daily activities, use of splints, tendon and nerve gliding exercises, ESWT, manual therapy, kinesiotaping, physical therapy agents, medical symptomatic treatments, injections into the carpal tunnel and surgical treatment options. .

Suspected risk factors for CTS include diabetes mellitus, menopause, hypothyroidism, obesity, arthritis, and pregnancy. Since hypothyroidism, menopause, and pregnancy are risk factors, there is a strong suspicion that hormonal changes may play a role in the etiology of CTS; however, no evidence was found to support this hypothesis.

In the diagnosis of CTS, a comprehensive and accurate clinical history should be taken together with the exclusion of other possible causes. The syndrome is characterized by intermittent and then increasing nocturnal paresthesia and dysesthesia findings. Later, sensory loss develops with hand muscle weakness and muscle atrophy of the thenar region, resulting from extensive axonal degeneration in the course of the disease. This set of symptoms is quite typical and rarely occurs in disorders other than CTS. In severe CTS cases, paresthesia symptoms may spread to the proximal forearm and upper arm, and sometimes to the shoulder(3).

In the following periods, loss of strength and atrophy of the thenar region muscles may occur. The diagnosis is made by clinical examination, electrophysiological methods (EMG) and imaging methods (such as ultrasound, magnetic resonance imaging). The clinical examination consists of sensory-motor examination and provocative tests. 1-2-3 on sensory examination. numbness with touch (paresthesia) or low sense of touch (hypoesthesia) in the fingers are detected. Motor examination may be normal in the early stage, and later on, weakness (weakness) in the thumb abducting and opposing muscle is detected.

In the first of the provocative tests, when the inside of the patient's wrist is hit with a reflex hammer, the patient usually feels an electric shock sensation in the first 3 fingers of the hand or a tingling sensation spreading to these fingers. This is known as Tinel's sign. In another clinical test, the patient is asked to flex both wrists (both wrists are flexed and the backs of both hands are touching each other) for 1 minute. In case of numbness and tingling spreading to the fingers, the test is considered positive (significant). , this is called the 'Phalen test'. Another diagnostic method, EMG, is performed by recording and evaluating electrical signals coming from nerves and muscles, using electricity and needles to diagnose nerve and muscle diseases. In CTS, a decrease in the conduction velocity of the median nerve is detected. In the diagnosis of CTS, the diagnosis is mostly made when the clinical picture and electrophysiological findings are evaluated well, but magnetic resonance imaging may be useful in some special cases (formations such as space-occupying tumors).

CTS treatment is divided into conservative and surgical. Conservative treatment methods include splinting (an assistive device worn on the body to relieve the nerve), exercise (sliding movements of the median nerve in the wrist and wrist flexor tendons), local corticosteroid injection (corticosteroid injection into the carpal tunnel), and ultrasound (deep with sound energy) from physical therapy applications. tissue heating), TENS (pain relief by applying controlled low-voltage electric current to the nervous system through the skin with electrodes placed on the skin), paraffin bath (immersion of the hand in a heated paraffin pool), ergonomic arrangements. Surgical treatment includes decompression of the nerve (4).

Virtual reality; It is defined as the use of interactive simulations created with computer hardware and software to offer users opportunities to enter environments that look and feel like real-world objects and events. With the feeling of being in that environment and the possibility of interacting with the environment, it differs from products such as video and television(5).

Virtual reality applications are grouped under 2 main headings as "immersive" and "non-immersive" according to the level of user coverage of the environment. The degree of inclusiveness of the offered virtual environment depends on the level of interaction, as well as the ability to isolate the user from stimuli outside the virtual environment (such as external sounds and lights). In immersive virtual reality systems, head-mounted screens (in the form of head-mounted display; headgear, mask or glasses) are used, while non-immersive virtual reality systems use screens(6). In this research the investigators aim to present the virtual reality-mediated exercise program to patients non-immersive. It is planned to use the Leap Motion motion sensor to detect hand and wrist movements and to monitor the gamified setup on the computer screen. The Leap Motion sensor is a hand motion sensor that rests on a stable platform and has no wearable or mountable parts on the patient. The Leap Motion sensor, whose main use is to control computers hands-free, has no potential harm to patients. Within the scope of this research, no part will be placed on the hand or wrist of the patients, they will only be asked to move their hands at a distance of 30 cm from the relevant sensor.

In the system that will be presented via computer and hand motion sensor, the patient will be asked to perform therapeutic exercises for the diagnosis of CTS in a scenario developed through virtual reality. The investigators predict that patients will actively participate in virtual reality-mediated therapeutic exercise program with high motivation and their functional results will be better than classical exercise programs.

The use of different rehabilitation protocols, which are also referred to as "serious games" in the medical field, in gamification and treatment has recently attracted attention. Virtual reality-mediated exercises are used for neurological rehabilitation to reduce disability caused by different neurological diseases such as cerebral palsy, stroke, Parkinson's Disease, multiple sclerosis, neurodegenerative diseases(7). In addition to neurological diseases, virtual reality-based rehabilitation methods; It has also been used in studies for scoliosis exercises, cardiac rehabilitation, chronic pain management, and pulmonary rehabilitation and its effectiveness has been demonstrated (8,9,10).

In our research, the investigators aim to present the tendon and nerve gliding exercises with proven effectiveness in patients with CTS, with non-immersive virtual reality systems, and to compare their effectiveness with the classical exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Having an EMG of the last 1 year and a diagnosis of mild and moderate CTS in this EMG,
* Between the ages of 20-70,
* Using a resting splint for the diagnosis of CTS,
* It was determined that he agreed to participate in the exercise program and to stop other therapeutic interventions to be applied to the wrist during the 3-month follow-up period.

Exclusion Criteria:

* Having a history of Cervical Radiculopathy,
* Having a diagnosis of rheumatoid arthritis,
* Having a history of acute trauma,
* Steroid injection to the wrist in the last 3 months,
* Having undergone wrist surgery in the last 3 months,
* Having an open wound around the wrist,
* Presence of uncontrolled disease (endocrinological, cardiovascular, pulmonary, hematological, hepatic, renal) was determined as patients with a history of active systemic inflammatory disease and/or malignancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Questionnaire | Change in this scale will be evaluated before the intervention, 1 month, and 3 months after the intervention.
  It is used to assess symptom severity and functional capacity in CTS. This scale is scored between 19-95 points, with higher scores indicating worse results.
Nerve conduction study | Change in this scale will be evaluated before the intervention, 1 month, and 3 months after the intervention
  It will be done to evaluate the involvement of the median nerve from CTS.
Median nerve area | Change in this scale will be evaluated before the intervention, 1 month, and 3 months after the intervention
  The median nerve area will be measured by ultrasound.
Visual Analog Scale | Change in this scale will be evaluated before the intervention, 1 month, and 3 months after the intervention
  Pain status will be evaluated with visual analog scale. This scale is scored between 0-10 points, with higher scores indicating worse results.
Hand grip strength | Change in this scale will be evaluated before the intervention, 1 month, and 3 months after the intervention
  The hand grip and pinch strength of the patients will be evaluated with a dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmet Kıvanç Menekşeoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not planned to share patient and study information with third parties.